CLINICAL TRIAL: NCT00385840
Title: A Study to Evaluate the Immunogenicity, Safety and Reactogenicity of a Second Vaccination With the Adjuvanted Influenza Vaccine Candidate Compared to Fluarix™ Administered Intramuscularly in Elderly Aged 60 Years and Above.
Brief Title: Study to Evaluate the Immunogenicity and Safety of a Second Vaccination With the Adjuvanted Influenza Vaccine Candidate
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 108708
Record Dates: First submitted 2006-10-10; First posted 2006-10-11 (Estimated); Results first posted 2013-04-29 (Estimated); Last update posted 2018-06-08 (Actual); Status verified 2016-10

CONDITIONS: Influenza
Keywords: Influenza vaccine; Influenza
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (2):
- Fluarix Group (Active Comparator): Subjects aged 60 years or older at the time of re-vaccination, who previously received 1 dose of the Fluarix™ vaccine in study NCT00321763, received 1 dose of Fluarix™ vaccine in this study. The vaccine was administered intramuscularly in the deltoid region of the non-dominant arm.
  Interventions: Biological: FluarixTM
- GSK1247446A Group (Experimental): Subjects aged 60 years or older at the time of re-vaccination, who previously received 1 dose of the GSK1247446A vaccine in study NCT00321763, received 1 dose of adjuvanted GSK1247446A vaccine in this study. The vaccine was administered intramuscularly in the deltoid region of the non-dominant arm.
  Interventions: Biological: Influenza Vaccine GSK1247446A

INTERVENTIONS:
Biological: Influenza Vaccine GSK1247446A — Single dose, intramuscular injection
  Arms: GSK1247446A Group
Biological: FluarixTM — Single dose, intramuscular injection
  Arms: Fluarix Group

SUMMARY:
The purpose of this study is to evaluate the immunogenicity and the safety of a second vaccination with candidate vaccine compared to Fluarix™ administered intramuscularly in elderly aged 60 years and above

DETAILED DESCRIPTION:
The Protocol Posting has been updated in order to comply with the FDA Amendment Act, Sep 2007.

ELIGIBILITY:
Inclusion Criteria:

* A male or female age 60 years or older at the time of the revaccination, who previously participated in 107192 & 107214 clinical trials.
* Subjects who the investigator believes can and will comply with the requirements of the protocol
* Written informed consent obtained from the subject.
* Free of an acute aggravation of the health status as established by clinical examination before entering into the study.

Exclusion Criteria:

* Use of any investigational or non-registered product (drug or vaccine) within 30 days preceding the administration of the study vaccine, or planned use during the study period.
* Acute clinically significant pulmonary, cardiovascular, hepatic or renal functional abnormality, as determined by physical examination or laboratory screening tests.
* Chronic administration (defined as more than 14 days) of immunosuppressants or other immune-modifying drugs within 3 months prior to the first vaccine dose.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination
* Administration of immunoglobulins and/or any blood products within the 3 months preceding the first dose of study vaccine or planned administration during the study period.
* Administration of other licensed vaccines within 2 weeks (for inactivated vaccines) or 4 weeks (for live vaccines) prior to enrolment in this study. Planned administration of a vaccine not foreseen by the study protocol up to 30 days after vaccination.
* History of hypersensitivity to a previous dose of influenza vaccine.
* History of confirmed influenza infection within the last 12 months.
* History of allergy or reactions likely to be exacerbated by any component of the vaccine(s)
* Acute disease at the time of enrolment.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 678 (Actual)
Dates: Start 2006-10-20; Primary Completion 2007-02-01 (Actual); Study Completion 2007-02-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (4):
- Norway (4):
  - GSK Investigational Site, Elverum
  - GSK Investigational Site, Hamar
  - GSK Investigational Site, Paradis
  - GSK Investigational Site, Stavanger

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Individual Participant Data Set: 108708 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 108708 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 108708 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 108708 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 108708 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 108708 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Fluarix Group | GSK1247446A Group
Started | 133 | 545
Completed | 129 | 531
Not Completed | 4 | 14
Not completed — Adverse Event | 1 | 1
Not completed — Lost to Follow-up | 3 | 13

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fluarix Group | GSK1247446A Group | Total
Number analyzed (Participants) | 133 | 545 | 678
Age, Continuous [Mean (Standard Deviation); unit: Years] | 68.1 (5.78) | 68.4 (5.95) | 68.3 (5.91)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 82 | 284 | 366
  Male | 51 | 261 | 312

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Any and Grade 3 Solicited Local Symptoms.
Description: Assessed solicited local symptoms were ecchymosis, pain, redness and swelling. Any = Incidence of a particular solicited local symptom regardless of intensity grade. Grade 3 pain = Pain that prevented normal everyday activity. Grade 3 redness/swelling/ecchymosis = Redness/swelling/ecchymosis above 50 millimeters (mm).
Time Frame: During the 7-day (Days 0-6) post-vaccination period
Population: The analysis was performed on the Total Vaccinated cohort, on all vaccinated subjects with the vaccine administration documented and symptom sheet completed.
Measure: Number; unit: subjects
Arm/Group | Fluarix Group | GSK1247446A Group
Number analyzed (Participants) | 131 | 542
subjects
  Any Ecchymosis | 2 | 14
  Grade 3 Ecchymosis | 0 | 1
  Any Pain | 27 | 282
  Grade 3 Pain | 0 | 0
  Any Redness | 28 | 245
  Grade 3 Redness | 4 | 102
  Any Swelling | 16 | 186
  Grade 3 Swelling | 2 | 56

2. Primary Outcome: Number of Subjects With Any, Grade 3 and Related Solicited General Symptoms.
Description: Assessed solicited general symptoms were arthralgia, fatigue, fever, headache, muscle aches and shivering. Any = Incidence of a particular solicited general symptom regardless of intensity grade or relationship with the study vaccination. Any Fever = Axillary temperature equal to or above (≥) 37.5 degrees Celsius (°C). Grade 3 symptom = Symptom that prevented normal activity. Grade 3 fever = Axillary temperature > 39.0°C. Related = Symptom considered by the investigator to have a causal relationship to study vaccination.
Time Frame: During the 7-day (Days 0-6) post-vaccination period
Population: as for outcome 1
Measure: Number; unit: subjects
Arm/Group | Fluarix Group | GSK1247446A Group
Number analyzed (Participants) | 131 | 542
subjects
  Any Arthralgia | 10 | 96
  Grade 3 Arthralgia | 0 | 3
  Related Arthralgia | 7 | 78
  Any Fatigue | 16 | 152
  Grade 3 Fatigue | 0 | 5
  Related Fatigue | 13 | 130
  Any Fever | 1 | 35
  Grade 3 Fever | 0 | 1
  Related Fever | 0 | 29
  Any Headache | 15 | 140
  Grade 3 Headache | 0 | 1
  Related Headache | 10 | 116
  Any Muscle aches | 12 | 179
  Grade 3 Muscle aches | 0 | 8
  Related Muscle aches | 6 | 154
  Any Shivering | 11 | 120
  Grade 3 Shivering | 0 | 12
  Related Shivering | 6 | 102

3. Primary Outcome: Number of Subjects With Any, Grade 3 and Related Unsolicited Adverse Events (AEs).
Description: Unsolicited AE covers any AE reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Any = Any unsolicited AE regardless of intensity or relationship to vaccination. Grade 3 = Unsolicited AE that prevented normal activity. Related = Unsolicited AE assessed by the investigator as causally related to the vaccination.
Time Frame: During the 30-day (Days 0-29) post vaccination period
Population: The analysis was performed on the Total Vaccinated cohort, which included all vaccinated subjects.
Measure: Number; unit: subjects
Arm/Group | Fluarix Group | GSK1247446A Group
Number analyzed (Participants) | 133 | 545
subjects
  Any unsolicited AE(s) | 31 | 121
  Grade 3 unsolicited AE(s) | 1 | 9
  Related unsolicited AE(s) | 4 | 34

4. Primary Outcome: Number of Subjects With Any and Related Serious Adverse Events (SAEs).
Description: SAEs assessed include medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization, result in disability/incapacity or are a congenital anomaly/birth defect in the offspring of a study subject. Any SAE = Occurrence of any SAE regardless of intensity grade or relation to vaccination Related = SAE considered by the investigator to have a causal relationship to study vaccination.
Time Frame: During the entire study period (from Day 0 to Day 29)
Population: The analysis was performed on the Total Vaccinated cohort, which included all vaccinated subjects.
Measure: Number; unit: subjects
Arm/Group | Fluarix Group | GSK1247446A Group
Number analyzed (Participants) | 133 | 545
subjects
  Any SAE(s) | 1 | 2
  Related SAE(s) | 0 | 0

5. Secondary Outcome: Titers for Serum Hemagglutination Inhibition (HI) Antibodies Against 3 Strains of Influenza Disease.
Description: Titers are presented as geometric mean titers (GMTs). The 3 influenza strains assessed were A/New Caledonia, A/Wisconsin and B/Malaysia. The seropositivity cut-off assay was 1:10.
Time Frame: At Day 0 and Day 21
Population: The analysis was performed on the According-To-Protocol (ATP) cohort, which included all evaluable subjects for whom data concerning immunogenicity outcome measures were available and for whom results were available for antibodies against at least one study vaccine antigen component.
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | Fluarix Group | GSK1247446A Group
Number analyzed (Participants) | 125 | 513
titers
  A/New Caledonia at Day 0 | 65.9 [54.4 to 79.9] | 61.8 [56.6 to 67.3]
  A/New Caledonia at Day 21 | 111.6 [94.3 to 132.2] | 114.4 [105.8 to 123.8]
  A/Wisconsin at Day 0 | 59.4 [46.2 to 76.4] | 82.0 [72.6 to 92.5]
  A/Wisconsin at Day 21 | 187.4 [151.2 to 232.1] | 370.0 [339.2 to 403.6]
  B/Malaysia at Day 0 | 100.2 [83.1 to 120.7] | 112.1 [101.7 to 123.6]
  B/Malaysia at Day 21 | 158.7 [132.6 to 189.9] | 232.4 [215.1 to 251.0]

6. Secondary Outcome: Number of Seroconverted Subjects Against 3 Strains of Influenza Disease.
Description: A seroconverted subject was defined as a vaccinated subject who had either a pre-vaccination titer <1:10 and a post-vaccination titer ≥1:40 or a pre-vaccination titer ≥1:10 and at least a four-fold increase in post-vaccination titer. The 3 influenza strains assessed were A/New Caledonia, A/Wisconsin and B/Malaysia.
Time Frame: At Day 21
Population: as for outcome 5
Measure: Number; unit: subjects
Arm/Group | Fluarix Group | GSK1247446A Group
Number analyzed (Participants) | 125 | 513
subjects
  A/New Caledonia | 21 | 78
  A/Wisconsin | 52 | 271
  B/Malaysia | 10 | 99

7. Secondary Outcome: Number of Seroprotected Subjects Against 3 Strains of Influenza Disease.
Description: A seroprotected subject was defined as a vaccinated subject who had a serum HI titer ≥ 1:40. The 3 influenza strains assessed were A/New Caledonia, A/Wisconsin and B/Malaysia.
Time Frame: At Day 0 and Day 21
Population: as for outcome 5
Measure: Number; unit: subjects
Arm/Group | Fluarix Group | GSK1247446A Group
Number analyzed (Participants) | 125 | 513
subjects
  A/New Caledonia at Day 0 | 100 | 381
  A/New Caledonia at Day 21 | 119 | 483
  A/Wisconsin at Day 0 | 81 | 397
  A/Wisconsin at Day 21 | 117 | 507
  B/Malaysia at Day 0 | 111 | 442
  B/Malaysia at Day 21 | 118 | 507

8. Secondary Outcome: Seroconversion Factor for Hemagglutination Inhibition (HI) Antibodies Against 3 Strains of Influenza Disease.
Description: The seroconversion factor (SCF) was defined as the fold increase in serum Hemagglutination Inhibition (HI) geometric mean titers (GMTs) post vaccination compared to Day 0. The 3 influenza strains assessed were A/New Caledonia, A/Wisconsin and B/Malaysia.
Time Frame: At Day 21
Population: as for outcome 5
Measure: Mean (95% Confidence Interval); unit: fold increase
Arm/Group | Fluarix Group | GSK1247446A Group
Number analyzed (Participants) | 125 | 513
fold increase
  A/New Caledonia | 1.7 [1.5 to 1.9] | 1.9 [1.8 to 2.0]
  A/Wisconsin | 3.2 [2.6 to 3.8] | 4.5 [4.1 to 5.0]
  B/Malaysia | 1.6 [1.4 to 1.7] | 2.1 [1.9 to 2.2]

ADVERSE EVENTS:
Time Frame: SAE(s): during the entire study period (Days 0-29); Solicited local and general symptoms: during the 7-day (Days 0-6) post-vaccination period; Unsolicited AE(s): during the 30-day (Days 0-29) post vaccination period.
Description: For the systematically assessed other non-serious AEs, the number of participants at risk included those from Total Vaccinated cohort whose symptom sheet had been completed.
Arm/Group | Fluarix Group | GSK1247446A Group
Serious Adverse Events (participants affected / at risk) | 1/133 | 2/545
Other Adverse Events (participants affected / at risk) | 66/133 | 434/545
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Fluarix Group (N=133) | GSK1247446A Group (N=545)
Cholelithiasis (Hepatobiliary disorders) | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 1
Pneumonia (Infections and infestations) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Sudden death (General disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Fluarix Group (N=133) | GSK1247446A Group (N=545)
Nasopharyngitis (Infections and infestations) | 13 | 33
Pain (General disorders) | 27/131 | 282/542
Redness (General disorders) | 28/131 | 245/542
Swelling (General disorders) | 16/131 | 186/542
Arthralgia (General disorders) | 10/131 | 96/542
Fatigue (General disorders) | 16/131 | 152/542
Fever (General disorders) | 1/131 | 35/542
Headache (General disorders) | 15/131 | 140/542
Muscle aches (General disorders) | 12/131 | 179/542
Shivering (General disorders) | 11/131 | 120/542

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.